CLINICAL TRIAL: NCT00541671
Title: Prevention of Narcotic-induced Nausea With Promethazine, a Randomized, Double-blind Placebo-controlled Trial
Brief Title: Prevention of Narcotic-Induced Nausea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated: recruiting or enrolling participants has halted prematurely and will not resume; participants are no longer being examined or treated
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 27002
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Results first posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Nausea
Keywords: Narcotics; Nausea
MeSH Terms: conditions — Nausea | interventions — Sodium Chloride; Promethazine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Patients will then be randomized to receive placebo, consisting of 10ml of normal saline solution to be administered intravenously with the narcotic
  Interventions: Drug: Saline
- 2 (Active Comparator): Patients will be randomized to 6.25mg of promethazine, consisting of 0.25ml of promethazine diluted in 9.75ml of normal saline.
  Interventions: Drug: Phenergan

INTERVENTIONS:
Drug: Saline — 10 c of saline
  Arms: 1
Drug: Phenergan — Physician ordered dose
  Arms: 2

SUMMARY:
We are doing this study to find out if extra medicine is needed to avoid the chance of nausea sometimes linked to narcotic pain medicine (for example, morphine, dilaudid, fentanyl). Some doctors always give medicine to prevent the possible side effect of nausea, while others do not. We are looking to see if this extra medicine is helpful in preventing nausea. The goal is to screen all patients with pain and enroll enough subjects to reach our goal of 164 evaluable study participants.

DETAILED DESCRIPTION:
Patients will be randomized to one of two study groups. They will then be asked to rate their pain and nausea on a line graph. If the patient is a female of child bearing age, a urine pregnancy test will be done per standard of care. After this, an IV catheter will be placed in a vein in the patients arm. Pain medicine will be given through this IV per the doctor's order. With this medicine, patients will be given 10 milliliters (2 teaspoons) of either Sodium Chloride (salt water) or Phenergan mixed with Sodium Chloride (salt water). Phenergan is a medication typically used to help with nausea and is a common ingredient in prescription cough medicine.

After this is finished, patients will be asked to rate their pain and nausea in 30 minutes, and again 1, 2, and 4 hours later. If the doctor decides the patient is able to be discharged from the emergency room before the 4 hours are up, they will be asked to rate your pain and nausea again before going home, and the study will be stopped at that time.

ELIGIBILITY:
Inclusion Criteria:

1. Patient in Christian Care Emergency Department
2. Require intravenous narcotics for painful condition
3. ≥18 years of age
4. Able to visually rate amount of pain and nausea

Exclusion Criteria:

1. Hypersensitivity to promethazine or opioids
2. Patient requesting anti-emetic at enrollment
3. Narcotic administration in last 6 hours
4. Pregnancy or currently breast-feeding
5. Known seizure disorder
6. Medical Instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perraut, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients will then be randomized to receive placebo, consisting of 10ml of normal saline solution to be administered intravenously with the narcotic
- Promethazine: Patients will be randomized to 6.25mg of promethazine, consisting of 0.25ml of promethazine diluted in 9.75ml of normal saline.
Period: Overall Study
Arm/Group | Placebo | Promethazine
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Not enough subjects were enrolled into this study. No analysis of data was performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Promethazine | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Customized [Number; unit: participants]
  Greater than or equal to 18 | 12 | 13 | 25
Sex/Gender, Customized [Number; unit: participants] | NA — Not collected because not relevant. | NA — Not Collected because not relevant. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Became Nauseated After IV Opiate Administration.
Time Frame: 4 hours post opiate administration
Measure: Number; unit: participants
Arm/Group | Placebo | Promethazine
Number analyzed (Participants) | 12 | 13
participants | 5 | 4

ADVERSE EVENTS:
Time Frame: Subjects were followed for 4 hours post drug/placebo administration.
Arm/Group | Placebo | Promethazine
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

LIMITATIONS AND CAVEATS:
Early termination due to small numbers of subjects and incomplete data for analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes